CLINICAL TRIAL: NCT00530244
Title: The Effect of Formula Fortified With Docosahexaenoic Acid (DHA) on Infants With Cystic Fibrosis (CF)
Brief Title: Use of Formula Fortified With DHA in Infants With Cystic Fibrosis
Acronym: DHA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Collaborators: Cystic Fibrosis Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: OSULLI03A0; H-10721 (Other: UMass Worcester)
Record Dates: First submitted 2007-09-13; First posted 2007-09-17 (Estimated); Last update posted 2018-03-07 (Actual); Status verified 2018-03

CONDITIONS: Cystic Fibrosis
Keywords: cystic fibrosis; fatty acids; docosahexaenoic acid; infant formula; growth; pancreatic function
MeSH Terms: conditions — Cystic Fibrosis | interventions — Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 1 (Experimental): Infants will be fed formula supplemented with docosahexaenoic acid
  Interventions: Dietary Supplement: Docosahexaenoic acid (DHA)
- 2 (Placebo Comparator): Infants will be fed standard formula (Enfamil)
  Interventions: Dietary Supplement: Standard formula (Enfamil)

INTERVENTIONS:
Dietary Supplement: Docosahexaenoic acid (DHA) — Infant formula with 0.96% of fatty acids as DHA
  Other Names: LIPIL x 3
  Arms: 1
Dietary Supplement: Standard formula (Enfamil) — This is a standard, commercially available infant formula.
  Other Names: Enfamil
  Arms: 2

SUMMARY:
The hypothesis of this study is that feeding infants diagnosed with CF via newborn screening a formula enhanced with a specific fish-oil fatty acid known as DHA will improve growth and decrease pancreatic dysfunction (as measured by human fecal elastase-1 in stool) over the first year of life.

Briefly, infants diagnosed with CF in the first month of life whose parents chose not to breast feed their babies will be invited to enroll in a study comparing a standard commercial infant formula (Enfamil) with a formula enriched with arachidonic acid (AA) and docosahexaenoic acid (DHA). The study formula has 3 times the amount of DHA available in commercially available formulas. Infants will have monthly tests of stool elastase and blood work at entry, 3, 6, 9 and 12 months of age.

DETAILED DESCRIPTION:
This study brings together several areas of CF and non-CF research: the finding that CF knock-out mice exhibit an abnormality in AA/DHA ratio in membrane bound fatty acids from tissue which expresses CFTR; the fact that very high doses of DHA fed to CF knock-out mice can correct many of the abnormalities seen in these animals; research on fatty acid content in human breast milk; the effects of breast feeding in CF; and the fact that newborn screening for CF is becoming more widespread and may allow for therapeutic interventions very early in life. This is the first study of which we are aware to look at a therapeutic intervention in children diagnosed with CF by newborn screening.

Fatty Acid Metabolism in CF It has been recognized for years that patients with CF have abnormalities in their fatty acid profile.(1) Initially, this was felt to be secondary to malabsorption of essential fats. However, in 1986, Strandvik's laboratory proposed that an abnormality in fatty acid turnover (specifically arachidonic acid metabolism) was a primary problem in patients with CF(2). More recently, Freedman et al (3) have shown that CFTR knockout mice have an abnormality in membrane bound long chain polyunsaturated fatty acids in CFTR expressing tissue with an increased ratio of arachidonic acid (AA) to docosahexanoic acid (DHA) compared to control animals. They have also shown that therapy with formula fortified with high doses of DHA reverses the lipid abnormality and ameliorates the pancreatic duct changes seen in these mice and decreases the inflammatory response to inhaled lipopolysaccharide(3,4).

Freedman et al (5) have gone on to show that abnormalities in membrane bound fatty acids in CFTR expressing tissues in humans are similar to that seen in CF knockout mice. They and Strandvik et al(6) have shown that this fatty acid abnormality is dependent on genotype with more severe fatty acid abnormalities found in patients with "severe" mutations (mutations associated with pancreatic insufficiency). That this abnormality is a primary part of the disease and not secondary to malabsorption is supported by the fact that obligate heterozygotes have fatty acid abnormalities intermediate between affected individuals and normal controls(5). In summary, fatty acid abnormalities appear to be a primary defect in CF and are directly related to the patient's genotype. Furthermore, dietary correction of this fatty acid imbalance improves symptoms in mice. Previous human studies looking at correction of fatty acid imbalances in CF patients have focused on the 18 carbon precursors to AA and DHA (reference 7, for example) or have used very brief treatment periods with eicosapentaenoic acid (EPA) (which was not effective in Freedman's mice) in individuals who already have established disease (8).

Human Breast Milk and Breast Feeding in CF Human breast milk contains low levels of DHA but standard infant formula does not (9).

Traditional infant formulas such as Similac and Enfamil have 18 carbon fatty acids as their source of long chain polyunsaturated fatty acids. These include linoleic acid (18 carbons, 2 double bonds, the last double bond 6 carbons from the methyl end; 18:2n-6) and linolenic acid (18:3n-3). Eighteen carbon fatty acids may be desaturated and elongated to make AA (20:4n-6) and DHA (22:6n-3) which are then incorporated into membrane phospholipids (10). Alternately, these 18 carbon fatty acids can be 0-oxidized in mitochondria and used as an energy source. AA and DHA are necessary for brain growth.(11) The most rapid period of brain growth is the third trimester and it seems likely that this is the most important period of time for accumulation of these fatty acids by the fetus. Prematurely born infants miss out on placental transfer of AA and DHA in the last trimester. They are also more likely to need to use long chain polyunsaturated fatty acids as an energy source since they may have limited caloric intake and increased caloric expenditure due to respiratory disease. It is not surprising, therefore, that AA and DHA supplemented formulas would be found to have a more profound effect upon pre-term than term infants. In fact, new formulas containing AA and DHA have been found to improve neurodevelopment in premature infants (12). However, there is controversy as to whether or not there are neurodevelopmental advantages to term infants being fed fatty acid supplemented formula with some authors reporting a benefit (13) and others (including a very large, double blind, randomized study(14) not finding any difference between term infants fed standard formula and those given long chain polyunsaturated fatty acid supplemented formula. Since brain tissue does not express CFTR and brain levels of AA and DHA were not abnormal in Freedman's mouse experiments (3), it seems unlikely that full term humans with CF would have neurodevelopmental problems related to decreased brain DHA levels different from the general population.

There is a limited reserve of n-3 fatty acids in tissues resulting in faster onset of DHA than AA depletion in infants who have a limited intake of fatty acids. This could be exaggerated in infants with CF in CFTR expressing tissue which is already low in DHA. Dietary AA and DHA are preferentially acylated into tissue structural lipids, whereas dietary 18 carbon n-3 and n-6 fatty acids can be more readily used as an energy source (10). Thus for some infants (premature infants and possibly CF infants) the longer chain fatty acids may be essential dietary components.

The 20 and 22 carbon n-3 fatty acids (EPA and DHA) inhibit 0-6 desaturase and reduce synthesis of AA from linoleic acid (18:2 n-6). (10) Therefore, unbalanced addition of DHA to infant diets may result in abnormal tissue fatty acid composition. Taking advantage of this desaturase inhibition by feeding infants a formula with DHA but without AA might be beneficial for infants with CF assuming that they have intrinsically elevated AA tissue levels and decreased DHA levels. However, such a strategy has not been tested and since there is a normal AA/DHA ratio in non-CFTR expressing tissues this strategy might put CF infants at risk of abnormal brain development by altering normal neural AA/DHA ratios. It seems prudent to provide both AA and DHA to CF infants in levels consistent with those found in human breast milk.

There is a great deal of variation in human breast milk long chain polyunsaturated fatty acid content depending on the mother's diet with DHA levels ranging from as little as 0.2% of fatty acids in women on vegetarian diets to 2.78% of fatty acids in Chinese women on a marine diet (9,15). DHA has been granted GRAS status ("generally recognized as safe") by the FDA, clearing its way for addition to infant formulas. Recently, Mead Johnson and Ross Laboratories have released infant formulas enriched with long chain polyunsaturated fatty acids, specifically AA and DHA. Many studies have demonstrated the safety of these formulas (13,14,16,17).

Given that breast milk contains low levels of DHA and traditional formula does not, it is reasonable to think that breast feeding might be beneficial for children with CF. Very few studies have looked at this question. In the 1960s and 1970s several authors warned against breast feeding because it was felt to precipitate hypoproteinemic, edematous states (18,19) By 1990 77% of CF Centers were recommending breast feeding for infants with CF (which means 23% were not). (20) In 1991 Holliday et al (21) were able to demonstrate improved growth in CF infants who were breast fed compared to those who were not. This study showed that breast feeding was safe for infants with CF and possibly beneficial.

A recent nationwide survey has demonstrated an association between breast feeding and improved outcome in CF individuals (22). Whether this is due to DHA, other constituents of breast milk not found in commercial formula, or social factors is not clear. Related to this survey result is the observation that some CFTR knockout mice do not develop pancreatic insufficiency and CF gastrointestinal symptoms until they are weaned from their mother's milk (Steven Freedman, personal communication). Mouse breast milk, like human milk, contains DHA. Although 15% of humans with CF are born with obvious pancreatic insufficiency and bowel obstruction (meconium ileus), many are not symptomatic on day one of life. Pancreatic insufficiency appears to be a continuous, not discrete, variable with change in pancreatic sufficiency status over time seen in many patients. In one study, only sixty percent of infants with CF diagnosed using newborn screening were noted to be pancreatic insufficient at diagnosis as determined by 72 hour fecal fat studies (23). By 12 months of age fat malabsorption was seen in 92% of this cohort. These results are similar to those of Waters et al (24) who also saw increasing prevalence of pancreatic dysfunction over time. It is speculated that early intervention with a DHA containing formula might slow the inflammatory destruction of the pancreas seen in humans over the first year of life.

LIPIL, manufactured by Mead Johnson has 0.32% fat as DHA. Mead Johnson has made a formula with three times this amount of DHA for this study. The study formula, designated LIPIL x 3, has 0.96% of fatty acids as DHA and retains the same AA concentration (0.64%) as the commercial formula. This formula meets the FDA GRAS designation and does not require an IND for use in a clinical trial.

Human infants have thrived for decades with the standard formulas that have been available; it remains unclear if term infants derive benefit from the long chain polyunsaturated fatty acids supplied by the newer formulas. Evidence indicates that term infants do well with either conventional or fatty acid supplemented formula so there is no ethical dilemma to a double-blind comparison of these formulas.

Newborn Screening for CF Many states have begun performing newborn screening for cystic fibrosis. For example, Massachusetts began screening for CF in February 1999. This program utilizes both IRT measurement and 39 mutation analysis. This has proved to be very good for detecting children with CF early in life, the median age at diagnosis being 16 days (Anne Commeau, personal communication). Many other states have begun performing newborn screening for CF using a similar algorithm or an IRT/IRT algorithm in which two blood samples are analyzed for IRT days apart. Compared to children diagnosed by conventional methods, Farrell et al (25,26) have shown improvement in the nutritional status of CF patients detected by newborn screening. It is believed that improved nutrition will lead to improved pulmonary function later in life, but to date this has not been proven. In fact, the finding that it is possible that newborn screening could lead to earlier acquisition of Pseudomonas aeruginosa has worried some clinicians about the utility of newborn screening for this disease (27,28). Thus, CF can be detected early in life using newborn screening and this has been shown to lead to nutritional and possibly pulmonary benefits over time.

It is the goal of this study to see if a simple intervention early in life in those children diagnosed with CF via newborn screening can make a difference in the progression of their disease. It is hypothesized that if humans respond to DHA in a similar fashion to CFTR knockout mice, then supplementation of these infants' diets with DHA early in life will provide protection from pancreatic disease and pulmonary inflammation.

ELIGIBILITY:
Inclusion Criteria:

* Infant diagnosed with CF and enrolled by 56 days of life
* Parental consent obtained

Exclusion Criteria:

* History of meconium ileus at birth that is resolved without surgical intervention (ie enema)
* History of bowel resection for any reason
* Breast feeding
* Premature birth (<34 weeks gestation)
* Severe cholestasis (Direct Bilirubin > 2x upper limit of normal for age)
* Severe hypoalbuminemia (Albumin < 2.5 gm/dl)

Max Age: 56 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 76 (Actual)
Dates: Start 2003-03; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
height and weight for age z-score and human fecal elastase-1 in stool | one year

SECONDARY OUTCOMES:
Secondary End Points: 1. AA/DHA ratio in plasma 2. Chest x-ray film Brasfield scores 3. Serum immune reactive trypsinogen 4. Serum alpha fetoprotein 5. Infant pulmonary function tests (subset analysis) 6. Bayley's scales of childhood development | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Brian P O'Sullivan, MD, Principal Investigator — University of Massachusetts, Worcester
Locations (24):
- United States (24):
  - UAB/CHS Cystic Fibrosis Center, Birmingham, Alabama
  - Emory Cystic Fibrosis Center, Atlanta, Georgia
  - Blank Children's Hospital, Des Moines, Iowa
  - Cystic Fibrosis Care & Teaching Center, Wichita, Kansas
  - Kosair Charities, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital, Boston, Massachusetts
  - Baystate Medical Center, Springfield, Massachusetts
  - UMass Memorial Healthcare, Worcester, Massachusetts
  - Children's Mercy Hospital, Kansas City, Missouri
  - Monmouth Medical Center, Long Branch, New Jersey
  - The Respiratory Center for Children, Morristown, New Jersey
  - Albany Medical Center, Albany, New York
  - Children's Hospital, Buffalo, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - Strong Memorial Hospital, Rochester, New York
  - Univesity Medical Center, Stony Brook, New York
  - SUNY Upstate Medical Center, Syracuse, New York
  - Children's Hospital at Westchester Medical Center, Valhalla, New York
  - Lewis H Walker CF Pulmonary Center, Akron, Ohio
  - Lewis H Walker Cystic Fibrosis Center Division of Pulmonary, Akron, Ohio
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Mountain State University, Morgantown, West Virginia

REFERENCES:
- [Background] Freedman SD, Katz MH, Parker EM, Laposata M, Urman MY, Alvarez JG. A membrane lipid imbalance plays a role in the phenotypic expression of cystic fibrosis in cftr(-/-) mice. Proc Natl Acad Sci U S A. 1999 Nov 23;96(24):13995-4000. doi: 10.1073/pnas.96.24.13995. PMID 10570187
- [Background] Freedman SD, Blanco PG, Zaman MM, Shea JC, Ollero M, Hopper IK, Weed DA, Gelrud A, Regan MM, Laposata M, Alvarez JG, O'Sullivan BP. Association of cystic fibrosis with abnormalities in fatty acid metabolism. N Engl J Med. 2004 Feb 5;350(6):560-9. doi: 10.1056/NEJMoa021218. PMID 14762183
- [Background] Parker EM, O'Sullivan BP, Shea JC, Regan MM, Freedman SD. Survey of breast-feeding practices and outcomes in the cystic fibrosis population. Pediatr Pulmonol. 2004 Apr;37(4):362-7. doi: 10.1002/ppul.10450. PMID 15022134
- [Background] Walkowiak J, Herzig KH, Strzykala K, Przyslawski J, Krawczynski M. Fecal elastase-1 is superior to fecal chymotrypsin in the assessment of pancreatic involvement in cystic fibrosis. Pediatrics. 2002 Jul;110(1 Pt 1):e7. doi: 10.1542/peds.110.1.e7. PMID 12093988
- [Derived] O'Sullivan BP, Baker D, Leung KG, Reed G, Baker SS, Borowitz D. Evolution of pancreatic function during the first year in infants with cystic fibrosis. J Pediatr. 2013 Apr;162(4):808-812.e1. doi: 10.1016/j.jpeds.2012.10.008. Epub 2012 Dec 11. PMID 23245194